CLINICAL TRIAL: NCT03423264
Title: A Phase II Randomized Trial of Prophylactic Gabapentin Plus Best Supportive Care Versus Best Supportive Care Alone for Patients Receiving Induction Chemotherapy Followed by Response-Stratified Locoregional Therapy for Locoregionally-Advanced, HPV-Related Oropharyngeal Cancer: An Optima II Secondary Study
Brief Title: PROGRESS Trial - Prophylactic Gabapentin for Relief of Symptoms and Improved Swallowing
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to accrue
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB17-1550
Record Dates: First submitted 2018-01-26; First posted 2018-02-06 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Oropharyngeal Cancer; HPV-Related Squamous Cell Carcinoma
Keywords: HPV-related oropharyngeal cancer; oropharyngeal cancer; HPV-related squamous cell carcinoma; prophylactic gabapentin; Optima II study
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Participants receiving radiation therapy as part of the OPTIMA II trial (NCT03107182) will be randomized to receive prophylactic gabapentin plus best supportive care versus best supportive care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Experimental): Participants randomized to this arm will receive gabapentin beginning on evening of the first day of radiation treatment at a dose of 600 mg. Gabapentin will continue to be taken twice a day (morning and evening) for the next 4 days of radiation treatment at increasing doses (up to 900 mg). Participants will continue to receive standard best supportive care medications as per their treating physician's recommendation.
  Interventions: Drug: Gabapentin
- Supportive Care Only (No Intervention): Participants will receive standard best supportive care medications as per their treating physician's recommendation.

INTERVENTIONS:
Drug: Gabapentin — Gabapentin taken as follows:
  Day 1 (evening): 600 mg Day 2 (morning): 600 mg Day 2 (evening): 600 mg Day 3 (morning): 600 mg Day 3 (evening): 900 mg Day 4 (morning): 900 mg Day 4 (evening): 900 mg Day 5 (morning): 900 mg Day 5 (noon): 900 mg Day 5 (evening): 900 mg
  Other Names: Neurontin
  Arms: Gabapentin

SUMMARY:
Enrollment is only available to patients enrolled on the Optima II study (NCT03107182).

The purpose of this trial is to compare rates of opioid use at completion of radiation for patients with Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 2 oral mucositis after receiving definitive nonoperative locoregional therapy with or without prophylactic gabapentin as part of best supportive care for locoregionally-advanced, HPV-related oropharyngeal cancer. Secondary purposes include comparison of total equivalent opioid dosage above baseline opioid use at end of treatment, quality of life metrics, swallowing function, feeding tube dependence, and protocol compliance in patients managed with best support care with or without prophylactic gabapentin. Rates of gabapentin-related side effects and discontinuation will also be investigated.

DETAILED DESCRIPTION:
Enrollment is only available to patients enrolled on the Optima II study (NCT03107182).

Primary objective: To compare rates of opioid requirement as a function of supportive care in patients experiencing CTCAE grade ≥2 oral mucositis at completion of radiation or chemoradiation as part of OPTIMA II

Secondary objectives: To compare total opioid equivalent dose above baseline opioid requirement at end of radiation, quality of life metrics, swallowing function, feeding-tube dependence, and protocol compliance in patients managed with best supportive care with or without prophylactic gabapentin. To investigate rates of gabapentin-related toxicity and discontinuation for patients treated on protocol.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment to OPTIMA II trial (NCT03107182)

Exclusion Criteria:

* Ineligible for enrollment to OPTIMA II trial (NCT03107182)
* Prior gabapentin therapy
* Creatinine clearance of < 45 mL/minute
* Documented intolerance, allergy, or hypersensitivity to gabapentin
* Hemodialysis or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Rate of opioid use at end of radiation treatment | 5 days
  Comparison of opioid use as part of best supportive care in patients with CTCAE grade ≥ 2 oral mucositis at the end of radiation treatment given as part of OPTIMA II study.

SECONDARY OUTCOMES:
Total opioid dosage during radiation treatment | 5 days
  Comparison of total opioid dosage given as part of best supportive care in patients with CTCAE grade ≥ 2 oral mucositis at the end of radiation treatment given as part of OPTIMA II study.
Differences in head and neck symptoms | 24 months
  Measured by changes in patient reported head and neck specific symptoms
Differences in overall quality of life | 24 months
  Measured by changes in patient reported symptoms
Differences in chemotherapy-induced peripheral neuropathy symptoms | 24 months
  Measured by patient reported symptoms
Swallowing Function | 12 weeks
  1. Normal
  2. Within functional limits: abnormal oral or pharyngeal stage but able to eat regular diet; no modifications or swallowing precautions
  3. Mild impairment: mild dysfunction in oral or pharyngeal stage, requires modified diet; no therapeutic swallowing precautions
  4. Mild-moderate impairment: mild dysfunction in oral and pharyngeal stage, requires modified diet and therapeutic swallowing precautions
  5. Moderate impairment: moderate dysfunction in oral or pharyngeal stage, aspiration noted on exam, requires modified diet and swallowing precautions
  6. Moderate-severe dysfunction: moderate dysfunction in oral or pharyngeal stage, aspiration noted on exam, requires modified diet and swallowing precautions; requires primary enteral feeding support
  7. Severe impairment: severe dysfunction with significant aspiration or inadequate oropharyngeal transit to esophagus, NPO, requires primary enteral feeding support
Feeding Tube Dependence | 24 months
  Assessment of rates of feeding tube dependence during and after radiation treatment
Treatment Delays | 7 weeks
  Determine rate of unplanned radiation treatment delays.
Side Effects | 13 weeks
  Determine rate of gabapentin related side effects as per CTCAE v4.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Haraf, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States